CLINICAL TRIAL: NCT04296591
Title: Relationship Between Fetal Right Heart Doppler Findings With Lamellar Body and Fetal Lung Maturity
Brief Title: This Study Was to Investigate the Efficacy of Fetal Right Heart Doppler Findings in Determination of Pulmonary Maturity
Status: Completed | Type: Observational
Sponsor: Karadeniz Technical University (Other)
Responsible Party: Principal Investigator, erhan hüseyin cömert, research asistant, Karadeniz Technical University
Other Study IDs: EComert
Record Dates: First submitted 2020-02-25; First posted 2020-03-05 (Actual); Last update posted 2020-03-05 (Actual); Status verified 2020-03

CONDITIONS: Preterm Birth; Prenatal Care Late; Preterm Labor
Keywords: LAMELLAR BODY; pulmonary maturation; doppler ultrasonography; fetal pulmonary artery
MeSH Terms: conditions — Premature Birth; Obstetric Labor, Premature

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 6 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- study group: The study group consisted of late preterm cases(34-37 weeks of gestation) and
  Interventions: Diagnostic Test: fetal heart doppler findings
- control group: the control group consisted of term cases (<37 weeks of gestation).
  Interventions: Diagnostic Test: fetal heart doppler findings

INTERVENTIONS:
Diagnostic Test: fetal heart doppler findings — Doppler data of main pulmonary artery and right pulmonary artery, mitral valve e/a wave ratio and lamellar body count were determined as the main research parameters. In both groups, fetal thorax and heart circumference ratio, mitral e/a wave ratio, right pulmonary artery and main pulmonary doppler indexes (PI, RI, S / D, AT / ET) were evaluated before cesarean section.
  Other Names: lamellar body count

SUMMARY:
Objective: The aim of this study was to investigate the efficacy of fetal right heart doppler findings in determination of pulmonary maturity.

Materials and Methods: Pregnant women refered to the Department of Obstetrics and Gynecology at Karadeniz Technical University were included in the study. Pregnant women with pregestational or gestational diabetes mellitus, morbid obesity, thyroid dysfunction and fetal abnormality aneuploidy were not included in the study. The study was planned on women with late preterm and term pregnancy. Late preterm cases between 34-37 weeks were included in study group and term cases over 37 weeks were in control group. The doppler findings of main pulmonary artery and right pulmonary artery, mitral valve e/a wave ratio and lamellar body count were determined as the main outcomes. During caesarean section, 5cc amniotic fluid was taken to measure lamellar bodies count. Perinatal results of patients were recorded. p<0.05 was considered as statistical significance.

DETAILED DESCRIPTION:
MATERIAL AND METHODS This study is a prospective clinical study and it was initiated after the approval of Karadeniz Technical University Faculty of Medicine Clinical Research Ethics Committee numbered 2017/88.

Between 2017-2019 years, pregnant women included in the study who admitted to the Department of Obstetrics and Gynecology at Karadeniz Technical University. The study was planned on cases who will undergo cesarean section over 34. week of gestation. They were not included in the study if pregnant women with pregestational or gestational diabetes mellitus, morbid obesity, thyroid dysfunction and fetal anomaly diagnosed aneuploidy or anomaly. Demographic data, ultrasonographic data and doppler parameters of all patients were recorded and evaluated prospectively. Informed consent was obtained from all participants prior to participation to work. Newborn results after birth were recorded.

Patients were divided into two groups. The study group consisted of late preterm cases (34-37 weeks of gestation) and the control group consisted of term cases (<37 weeks of gestation).

Doppler data of main pulmonary artery and right pulmonary artery, mitral valve e/a wave ratio and lamellar body count were determined as the main research parameters. In both groups, fetal thorax and heart circumference ratio, mitral e/a wave ratio, right pulmonary artery and main pulmonary doppler indexes (PI, RI, S / D, AT / ET) were evaluated before cesarean section. All ultrasonographic examinations and measurements were performed by a single operator with color doppler ultrasonography device. Doppler measurements were performed in supine and slightly left-facing position. Doppler index measurements of two groups were recorded separately for each pregnant.

Lamellar Body Count Lamellar body counting; at least 2cc of amniotic fluid not infected with blood during the cesarean section was taken into the EDTA tube and not centrifuged in thestudy. The sample was studied by using automatic blood counting device which is used for counting the shaped elements of blood called Coulter Counter which makes automatic blood count in hematology laboratories. The value specified in the platelet count part was accepted as the number of lamellar bodies in the report.

Statistical analysis All data were analyzed using with IBM SPSS Statistics 11 (IBM SPSS, Turkey). In addition to descriptive statistical methods, Student's t test was used to compare the quantitative data.

ELIGIBILITY:
Inclusion Criteria:

* preterm and term pregnancy
* caesarean cases

Exclusion Criteria:

* pregestational diabetes mellitus
* gestational diabetes mellitus
* morbid obesity
* thyroid dysfunction
* fetal anomaly diagnosed an euploidy or anomaly.

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Gender Based: Yes — pregnancy woman
Study Population: total of 70 pregnant women (n: 70), 25 in the study group and 45 in the control group
Sampling Method: Non-Probability Sample
Enrollment: 1 (Actual)
Dates: Start 2017-01-01 (Actual); Primary Completion 2019-06-01 (Actual); Study Completion 2019-08-01 (Actual)

PRIMARY OUTCOMES:
lamellar body count | immediately after the procedure(1year)
  lamellar body count was higher in the control group
Doppler data of main pulmonary artery and right pulmonary artery, mitral valve e/a wave ratio | immediately after the procedure (1year)
  this data was measured before cesarian section.significant/ nonsignificant differences were detected between groups

CONTACTS AND LOCATIONS:
Overall Officials: ERHAN HUSEYIN COMERT, Principal Investigator — Karadeniz Technical University; TURHAN ARAN, PROF, Study Director — Karadeniz Technical University

IPD SHARING:
Plan to Share IPD: Undecided